CLINICAL TRIAL: NCT06938711
Title: A Rollover Protocol of Elacestrant, in Combination With Onapristone, for Patients With Estrogen Receptor-Positive, Progesterone Receptor-Positive, HER2-negative Advanced or Metastatic Breast Cancer
Brief Title: A Rollover Protocol of Elacestrant, in Combination With Onapristone, for Patients With ER+, PR+, HER2- Advanced or Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change in corporate strategy.
Sponsor: Context Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONA-XR-104
Record Dates: First submitted 2023-05-30; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant; RAD1901; onapristone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Elacestrant / Onapristone (Experimental): Elacestrant and Onapristone combination
  Interventions: Drug: Elacestrant; Drug: Onapristone

INTERVENTIONS:
Drug: Elacestrant — Elacestrant 200mg once daily oral dosing in cycles of 28 days.
  Other Names: RAD1901
Drug: Onapristone — Onapristone 40mg twice daily oral dosing in cycles of 28 days.

SUMMARY:
This is a rollover study for patients enrolled in the discontinued ELONA clinical trial (ONA-XR-103) with the primary objective to characterize the safety of elacestrant in combination with onapristone either alone or in combination.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently enrolled in the ELONA clinical study (ONA-XR-103) and receiving onapristone or elacestrant, either alone or in combination.
* Patient is currently benefiting from the treatment in the ELONA clinical study, as determined by the investigator.
* Patient currently has no evidence of progressive disease, as determined by the investigator.

Exclusion Criteria:

* Pregnant or nursing (lactating) women.
* Female patients of childbearing potential (e.g., are menstruating) who do not agree to abstinence or, if sexually active, do not agree to the use of highly effective contraception, throughout the study and for up to 30 days after stopping study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Characterize the safety of elacestrant in combination with onapristone. | 7 months
  Monitor the treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States